CLINICAL TRIAL: NCT00679900
Title: Comparison of the Safety and Efficacy of Eplivanserin and Lormetazepam in the Treatment of Insomnia Characterized by Sleep Maintenance Difficulties. A 4 Week, Randomized, Double-blind,Comparative, Parallel-group Study
Brief Title: Comparison of Eplivanserin and Lormetazepam in the Treatment of Insomnia Characterized by Sleep Maintenance Difficulties
Acronym: DREAMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD study director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10480; EudraCT 2007-003822-28
Record Dates: First submitted 2008-05-07; First posted 2008-05-19 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Primary Insomnia; Sleep Maintenance Difficulties
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — SR 46349B; lormetazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: eplivanserin (SR46349)
- 2 (Active Comparator)
  Interventions: Drug: lormetazepam

INTERVENTIONS:
Drug: eplivanserin (SR46349) — 5 mg/day
  Arms: 1
Drug: lormetazepam — 1 mg/day
  Arms: 2

SUMMARY:
The primary objective is to compare the potential for next-day residual effects of eplivanserin 5 mg/day and lormetazepam 1 mg/day by measuring the sleepiness in the morning using the patient's sleep questionnaire during 4 weeks of treatment in patients with chronic primary insomnia and sleep maintenance difficulties.

The secondary objectives are to compare the clinical safety of both products, including the potential for rebound insomnia and withdrawal symptoms after treatment discontinuation, to compare the efficacy of both products on subjective sleep parameters and to compare the effects of both products on patient's daytime functioning.

ELIGIBILITY:
Inclusion Criteria:

* Primary Insomnia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria
* At least 1 hour of wakefulness for at least 3 nights per week during the month preceding inclusion
* Disturbances of sleep maintenance criteria based on the patient's sleep questionnaire during the run-in period

Exclusion Criteria:

* Pregnant or breastfeeding women and women of childbearing potential without effective contraceptive method of birth control
* Night shift workers and individuals who nap 3 or more times per week
* Consumption of xanthine-containing beverages (i.e., tea, coffee or cola) that comprises more than 5 cups or glasses per day
* Insomnia secondary to a general medical condition

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Sleepiness in the morning measured on a visual analog scale of the patient's sleep questionnaire | 4 weeks

SECONDARY OUTCOMES:
Other measure of next-day residual effects (ability to concentrate of the patient's sleep questionnaire) | 4 weeks
Rebound effect measured by pr-WASO and pr-SOL on patient's sleep questionnaire during the run-out period | 4 weeks
Subjective sleep parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Barcelona, Spain